CLINICAL TRIAL: NCT02975830
Title: Tracheobronchial Angle in Children - Three-dimensional Computed Tomography Based Measurements
Status: Completed | Type: Observational
Sponsor: King Fahad Medical City (Other Government)
Responsible Party: Principal Investigator, Tariq Wani, Consultant Anesthesiologist, King Fahad Medical City
Other Study IDs: H-01-R-012/16-460
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Bronchus; Pediatric Airway

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 0-2 years: Children aged from birth to 24 months Three dimensional CT based images
  Interventions: Radiation: Three dimensional CT based images
- 2-4 Years: Children aged from 25-48 months Three dimensional CT based images
  Interventions: Radiation: Three dimensional CT based images
- 4-6 Years: Children aged from 49-72 Three dimensional CT based images
  Interventions: Radiation: Three dimensional CT based images
- 6-8 years: Children aged from 73-96 months Three dimensional CT based images
  Interventions: Radiation: Three dimensional CT based images

INTERVENTIONS:
Radiation: Three dimensional CT based images — Right bronchial angle, left bronchial angle

SUMMARY:
Accurate understanding of tracheobronchial anatomy is important for application of various airway maneuvers in anesthesiology in children. Majority of pediatric anesthesia textbooks state that the anatomic orientation of the right main bronchus is at less acute angle to the vertical tracheal axis, although these angles tend to be similar in children younger than three years of ageThe visualization of the air column in tracheobronchial tree in a three-dimensional (3D) CT-based image is clear with the air column simulating the actual internal shape of the airway.

We hypothesize that RBA and LBA are unequal as children like adults are prone to right mainstem intubation We have measured the right and left bronchial angle using the three dimensional CT based images of the air column in the tracheobronchial tree.

DETAILED DESCRIPTION:
Accurate understanding of tracheobronchial anatomy is important for application of various airway maneuvers in anesthesiology in children.

Significant variations and discrepancies in the reported tracheobronchial angles are found in literature.

Various imaging modalities ranging from chest x-ray to helical computed tomography (CT) have been used for measuring the tracheobronchial angles in children and the results are varied with some studies reporting equal angles [2016] while others reporting right bronchial angle to be smaller than left bronchial angle [Kubota].

The visualization of the air column in tracheobronchial tree in a three-dimensional (3D) CT-based image is clear with the air column simulating the actual internal shape of the airway. The highest quality medical-grade (3D) images are obtained using CT data [Uchida M]. Computed tomography (CT) is considered the current gold standard for airway measurements as the air-tissue interface is better delineated by CT imaging [Reinhardt].

We hypothesize that RBA and LBA are unequal as children like adults are prone to right mainstem intubation We have measured the right and left bronchial angle using the three dimensional CT based images of the air column in the tracheobronchial tree.

ELIGIBILITY:
Inclusion Criteria:

* CT scans airways

Exclusion Criteria:

* any disease that is anticipated to distort the normal shape of airways wee excluded from the study

Max Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: upto 8years of age
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
tracheobronchial angles | 6 months

IPD SHARING:
Plan to Share IPD: No